CLINICAL TRIAL: NCT00603005
Title: Adherence Improvement in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Dr. H.J.M. Beckers, MD, phD, Department of Ophthalmology, University Hospital Maastricht
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: MEC 07-1-015; CTCM-071015
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Glaucoma
Keywords: Glaucoma; Adherence
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Device: Use of TravAlert dosing aid with or without drop guider
- 2 (Experimental)
  Interventions: Device: Use of TravAlert dosing aid with or without drop guider
- 3 (Experimental)
  Interventions: Device: Use of TravAlert dosing aid with or without drop guider
- 4 (Experimental)
  Interventions: Device: Use of TravAlert dosing aid with or without drop guider

INTERVENTIONS:
Device: Use of TravAlert dosing aid with or without drop guider — Each patient will use a dosing aid and/or drop guider for 6 months

SUMMARY:
The purpose of this study is to study the effect on intraocular pressure in glaucoma patients using the TravAlert dosing aid with or without the Eyot drop guider and with or without additional patient education.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis glaucoma or ocular hypertension
* Treatment with travoprost or travoprost/timolol

Exclusion Criteria:

* High risk of side effects expected from travoprost or travoprost/timolol
* Absolute inability to administer eye drops
* Difficulty in reading or speaking Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 6 months

SECONDARY OUTCOMES:
Information with regard to the use of eye drops from data generated by the TravAlert dosing system | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Helena J Beckers, MD/phD, Principal Investigator — Maastricht University Medical Center
Locations (14):
- Netherlands (14):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - Medisch centrum Alkmaar, Alkmaar
  - Wilhelmina ziekenhuis, Assen
  - Amphia ziekenhuis, Breda
  - Deventer ziekenhuis, Deventer
  - Catharina ziekenhuis, Eindhoven
  - Groene hart ziekenhuis, Gouda
  - ziekenhuis de Tjongerschans, Heerenveen
  - Atrium medisch centrum, Heerlen
  - Westfries gasthuis, Hoorn
  - University hospital, Maastricht
  - Canisius Wilhelmina ziekenhuis, Nijmegen
  - Erasmus medisch centrum, Rotterdam
  - Isala klinieken, Zwolle